CLINICAL TRIAL: NCT06137391
Title: Effectiveness of Partial Pulpotomy and Pulpotomy in Symptomatic Deeply Carious Permanent First Molars With Molar Incisor Hypomineralisation (24 Months Randomised Controlled Clinical Trial)
Brief Title: Effectiveness of Pulpotomy in Carious First Permanent Molar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rodaina Helmy, Assistant Lecturer, Pediatric dentistry department, Faculty of dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0775-09/2023
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization | interventions — Apexification; Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIH and irreversible pulpitis (Experimental): Group I (n=48) diagnosed with MIH and irreversible pulpitis. Group I will be randomly equally allocated into Group I A (n=24): partial pulpotomy (PP) and Group I B (n=24): full pulpotomy (FP). If pulpal bleeding cannot be controlled within 6 minutes using cotton pellets soaked in 3% sodium hypochlorite, the allocated procedure will be abandoned. The pulpotomy agent to be used will be mineral trioxide aggregate (MTA) and teeth will be restored using a resin modified glass ionomer restoration (RMGIC).
  Interventions: Procedure: Vital Pulp Therapy
- No MIH with irreversible pulpitis (Active Comparator): Group II (n=48) diagnosed with irreversible pulpitis but not affected with MIH. Group II will be randomly equally allocated into Group II A (n=24): partial pulpotomy (PP) and Group II B (n=24): full pulpotomy (FP). If pulpal bleeding cannot be controlled within 6 minutes using cotton pellets soaked in 3% sodium hypochlorite, the allocated procedure will be abandoned. The pulpotomy agent to be used will be mineral trioxide aggregate (MTA) and teeth will be restored using a resin modified glass ionomer restoration (RMGIC).
  Interventions: Procedure: Vital Pulp Therapy

INTERVENTIONS:
Procedure: Vital Pulp Therapy — The pulp is accessed after caries removal then the inflamed part of the pulp is excavated. After haemostasis is achieved, a pulpootmy medicament is used to coronally seal the remaining pulp tissue. In partial pulpotomy only part of the pulp chamber is excavated while in full pulpotomy the whole pulp chamber is excavated.
  Other Names: Apexogenesis, Pulpotomy, Partial Pulpotomy

SUMMARY:
Pediatric dentists frequently encounter deeply carious young permanent first molars (PFM) with Molar Incisor Hypomineralisation (MIH). Pulpal status of affected PFM was found to be different from that of unaffected PFMs which consequently might influence the pulpal response after vital pulp therapy.

The aim of this study is to evaluate the clinical and radiographic effectiveness of partial removal of pulp in deeply carious symptomatic PFM affected with MIH over 24 months.

DETAILED DESCRIPTION:
Pediatric dentists frequently encounter deeply carious young permanent first molars (PFM) with Molar Incisor Hypomineralisation (MIH). Pulpal status of affected PFM was found to be different from that of unaffected PFMs which consequently might influence the pulpal response after vital pulp therapy. The aim of this study is to evaluate the clinical and radiographic effectiveness of partial removal of pulp in deeply carious symptomatic PFM affected with MIH over 24 months. In this prospective randomized controlled clinical trial, a randomized assigned sample of 96 children each with a deeply carious young PFM, Group I (n=48) diagnosed with MIH and irreversible pulpitis and Group II (n=48) diagnosed with irreversible pulpitis but not affected with MIH. Group I will be randomly equally allocated into Group II A (n=24): partial pulpotomy (PP) and Group I B (n=24): full pulpotomy (FP). Group II will also be randomly equally allocated into Group II A (n=24): PP and Group II B (n=24): FP. If pulpal bleeding cannot be controlled within 6 minutes using cotton pellets soaked in 3% sodium hypochlorite, the allocated procedure will be abandoned. The pulpotomy agent to be used will be mineral trioxide aggregate (MTA) and teeth will be restored using a resin modified glass ionomer restoration (RMGIC). Teeth will be followed up clinically and radiographically using periapical x-rays for 24 months. Cone beam computed tomographic scans will be taken initially and at 24 months. Pain levels will be scored preoperatively before local anesthetic administration and postoperatively every 24 hours for 7 days using visual analogue scale. All data will be statistically analyzed and discussed considering the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* 7-13-year-old children.
* At least one deeply decayed first permanent molar, checked through periapical x-ray)
* Noncontributory medical history.
* The tooth should be showing irreversible pulpitis signs and symptoms.
* The tooth is restorable and probing pocket depth and mobility within normal limits.
* No signs of pulpal necrosis including sinus tract or swelling.

Exclusion Criteria:

* Non-restorable teeth.
* Negative response to cold testing.
* Presence of sinus tract or swelling.
* No pulp exposure after caries excavation.
* Bleeding could not be controlled after partial pulpotomy in 6 minutes.
* Insufficient bleeding after pulp exposure; the pulp is judged necrotic or partially necrotic.
* History of analgesic intake 3 days prior to the day of commencement of procedure.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  Pain levels will be scored preoperatively before local anesthetic administration and postoperatively every 24 hours for 7 days using visual analogue scale, with 0 representing no pain and 100 representing pain as bad as it could be
Digitalized periapical Radiographs | Day 0, then at 6, 12, 18 and 24 months.
  Standardized digitalized periapical radiographs will be taken.
Cone Beam Computed Tomography scans | Day 0, 24 months
  Cone Beam Computed Tomography scans will be taken initially and at 24 months only to avoid excessive radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Rodaina H. Helmy, Principal Investigator — AlexU

IPD SHARING:
Plan to Share IPD: No